CLINICAL TRIAL: NCT02329041
Title: A Randomised Controlled Trial Comparing of McGrath Series 5 and Airtraq Videolaryngoscope for Double-lumen Tube Intubation in Patients With Low Airway Risk Index Score
Brief Title: Comparison of McGrath Series 5 and Airtraq Videolaryngoscope for Double-lumen Tube (DLT) Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wenlong Yao, M.D., Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJMZK201412002
Record Dates: First submitted 2014-12-21; First posted 2014-12-31 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Intubation;Difficult; Thoracic Disease; Intubation Complication
Keywords: videolaryngoscope; double-lumen tube; intubation
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- McGrath Series 5 (Experimental): DLT intubation with McGrath Series 5 videolaryngoscope
  Interventions: Device: McGrath Series 5
- Airtraq (Active Comparator): DLT intubation with Airtraq videolaryngoscope
  Interventions: Device: Airtraq

INTERVENTIONS:
Device: McGrath Series 5 — one kind of videolaryngoscopes, which are widely used in airway management.
  Arms: McGrath Series 5
Device: Airtraq — another kind of videolaryngoscopes, which are also widely used in airway management.
  Arms: Airtraq

SUMMARY:
Previous study showed that McGrath Series 5 videolaryngoscope is an alternative tool for double-lumen tube intubation. We have compared it with traditional Macintosh laryngoscopefor double-lumen tube intubation. In this study, we will investigate its role in double-lumen tube intubation by comparison with another videolarygoscope.

DETAILED DESCRIPTION:
The investigators designed a randomised controlled study to compare of McGrath Series 5 and Airtraq videolaryngoscope for DLT intubation in intubation time and the first attempt success rate.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Thoracic surgery required one lung ventilation

Exclusion Criteria:

* ASA physical status >4
* Emergent operation
* planned tracheotomy
* difficult intubation predicted by a simplified airway risk index score

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Intubation time | at intubation
  defined as time from inserting blade to mouth to withdrawal of blade, measured with a stopwatch

SECONDARY OUTCOMES:
number of successful intubation at first attempt | at intubation
total successful rate of DLT intubation | at intubation

OTHER OUTCOMES:
Airway evaluation with Cormack-Lehane Score | At intubation
  based on Cormack-Lehane classification. degree 1 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Yuke Tian, M.D., Study Chair — yktian@tjh.tjmu.edu.cn
Locations (1):
- Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Because the article has not been published.